CLINICAL TRIAL: NCT00512343
Title: Establishment of a Bank of Synovial Fluids and Paired Sera From Arthritic Patients for the Evaluation of New Methods Facilitating the Diagnosis and the Monitoring of Progression and Therapy of Arthritis.
Brief Title: Synovial Fluid Bank From Arthritic Patients
Status: Recruiting | Type: Observational
Sponsor: Gilles Boire (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Sponsor-Investigator, Gilles Boire, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: 02-12 LS
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Arthritis
Keywords: Synovial Fluid; Arthritis; Paired serum/synovial fluid samples
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluids from joints with effusion Sereum samples drawn on the same day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives of this group project is to collect synovial fluid (SF) and paired sera and carry out preclinical studies to evaluate, alone or by combination testings, the potential of novel biomarkers for their prevalence and diagnostic/prognostic values in patients with arthritis, and to determine how therapeutic intervention regulate their levels.

DETAILED DESCRIPTION:
Our group has developed interdisciplinary expertise in biomarkers related to distinct aspects of inflammation-induced joint damage, most notably those associated with degradation of components of the extracellular matrix, bone loss, or associated with post-translational changes on protease inhibitors.

The objectives of this group project is to collect SF and paired sera and carry out preclinical studies to evaluate, alone or by combination testings, the potential of novel biomarkers for their prevalence and diagnostic/prognostic values in patients with arthritis, and to determine how therapeutic intervention regulate their levels.

More specifically, we will study (1) biomarkers associated with osteoclastic bone resorption and synthesis/degradation of cartilage, (2) inhibitors of enzymes (calpastatin) that are preferentially targeted by rheumatoid patients, as well as (3) enzymes (e.g. Matrix Metalloproteinases (MMPs)) responsible for the cleavage of components of the articular cartilage.

Finally, we propose to characterize the repertoire of specific active proteases in the SF of arthritic patients concomitantly to the use biomarkers (neoepitopes of cleaved collagens) previously associated with cartilage destruction and synthesis to identify new targets for the development of protease inhibitors for the treatment of arthritis. Furthermore, our project will also provide the opportunity to test the potential of measuring the net proteolytic activity by Fluorescent-Activated Substrate Conversion as a method of monitoring disease activity and treatment efficiency in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Significant joint effusion

Exclusion Criteria:

* Hemorrhagic effusion
* Traumatic effusion
* Less than 3 ml total of collected fluid (used for routine analysis and culture)
* Inability or refusal to consent

Ages: 3 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suffering from various arthritides (rheumatoid arthritis, gout and other microcristalline arthritides, osteoarthritis, spondylarthropathies, juvenile idiopathic arthritis, and various other diseases, including inflammatory polyarthritis of recent-onset in adults
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2002-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Availability of paired synovial fluid and serum samples for exploratory studies | Use with various collaborators at different times, upon request and approbation
  Availability of paired synovial fluid and serum samples, linked with anonymized clinical and treatment data, from patients suffering from various arthritides (rheumatoid arthritis, gout and other microcrystalline arthritides, osteoarthritis, spondylarthropathies, juvenile idiopathic arthritis, and various other diseases, including inflammatory polyarthritis of recent-onset in adults

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boire, MD, MSc, Principal Investigator — CHUS and Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kilani RT, Maksymowych WP, Aitken A, Boire G, St-Pierre Y, Li Y, Ghahary A. Detection of high levels of 2 specific isoforms of 14-3-3 proteins in synovial fluid from patients with joint inflammation. J Rheumatol. 2007 Aug;34(8):1650-7. Epub 2007 Jul 1. PMID 17611984
- [Result] Simard N, Boire G, de Brum-Fernandes AJ, St-Pierre Y. A novel approach to measure the contribution of matrix metalloproteinase in the overall net proteolytic activity present in synovial fluids of patients with arthritis. Arthritis Res Ther. 2006;8(4):R125. doi: 10.1186/ar2014. PMID 16859524